CLINICAL TRIAL: NCT05713409
Title: Prediction and Close Monitoring of Postoperative Recurrence by Using Intestinal Ultrasonography After Ileocecal Resection in Crohn's Disease Patients
Brief Title: Prediction and Close Monitoring of Postoperative Recurrence by Intestinal Ultrasound After Ileocecal Resection in Crohn's Disease Patients
Acronym: INSIGHT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Krisztina Gecse, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_405 # 21.452
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with an established diagnosis of CD going through ileocecal resection
  Interventions: Diagnostic Test: Intestinal ultrasound

INTERVENTIONS:
Diagnostic Test: Intestinal ultrasound — As part of the routine care, patients will undergo ileocolonoscopy at 6 months, IUS will be performed 3, 6, 12, 18, 24, 30 and 36 months (using B-mode and CDS) and at 3 and 6 months elastography will be performed on the neo-terminal ileum. Biomarkers (CRP and fecal calprotectine) will be measured according to routine care.

SUMMARY:
Crohn's disease (CD) is an inflammatory bowel disease causing chronic transmural inflammation followed by intestinal complications including strictures and penetrating lesions such as fistulas and abscesses. 30-50% of the CD patients will require surgery during the course of their disease. Unfortunately, resection is not curative and endoscopically recurrent lesions (i.e. endoscopic recurrence) are observed in 65-90% of patients within 12 months, and in 80-100% within 3 years after the operation. Eventually 15-20% of patients will require new surgery within 5 years. Close monitoring for postoperative recurrence is therefore needed to perform early intervention and prevent clinical recurrence and need for re-surgery. Endoscopy is the gold standard to assess postoperative disease recurrence however it's limited by its invasiveness. Cross sectional imaging is known for accurate detection of postoperative recurrence. Intestinal ultrasound (IUS) of the colon and (neo)terminal ileum correlates well with CT, MRE and colonoscopy findings in the postoperative setting. IUS is non-invasive, cheap, readily available and may show early, signs of disease recurrence. Therefore it could be a useful tool to predict endoscopic recurrence at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Crohn's disease
* undergoing ICR (or re-resection)
* ≥16 years of age

Exclusion Criteria:

* <16 years of age
* Inability to give informed consent
* Ongoing gastroenteritis
* Deviating stoma
* (Sub)total colectomy
* Obesity (BMI >35 kg/m²)
* Insufficient visualization of the anastomosis AND the neo-terminal ileum at baseline IUS

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with established Crohn's disease going through ICR will be eligible for inclusion
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary aim of the study is to investigate if IUS (as measured by B-mode and CDS) in combination with faecal calprotectin at 3 months after ICR is an early surrogate marker of endoscopic disease recurrence (as defined by a RS ≥ i2) at 6 months | 6 months

SECONDARY OUTCOMES:
• To assess if IUS (as measured by B-mode, CDS and SWE) alone at 3 months after ICR is an early surrogate marker of endoscopic disease recurrence (as defined by a RS ≥ i2) at 6 months | 6 months
to assess if IUS (as measured by B-mode, CDS and SWE) alone or in combination with faecal calprotectin at 6 months after ICR is accurate in detecting endoscopic recurrence at 6 months (as defined by a RS score ≥ i2 and by the SES-CD˃3) | 6 months
to develop an IUS score for postoperative recurrence in Crohn's disease | 6 months
to assess if IUS (as measured by B-mode, CDS and SWE) alone or in combination with faecal calprotectin at 12 months after ICR is a surrogate marker of endoscopic disease recurrence (RS≥ 2) at 18 months and/or clinical outcomes at 18, 24, 30 and 36 months | 12-36 months
to compare IUS (as measured by B-mode, CDS and SWE; alone or in combination with faecal calprotectin) and the RS upon endoscopy at 6 months after ICR for their prognostic role on clinical outcomes upon 3 years of follow-up | 6 - 36 months
to assess if SWE during IUS at 3, 6 and 12 months is predictive of anastomotic stenosis upon follow-up | 3-12 months
to assess the feasibility of IUS in the postoperative settings for different types of anastomosis | 3-6 months
to assess the diagnostic accuracy of FCal at 3 and 6 months to predict and determine endoscopic disease recurrence, respectively | 3-6 months

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Klinikum Lüneburg, Lüneburg
  - Hospital of Oldenburg, Oldenburg
- Instituto Clinico Humanitas IRCSS, Milan, Rozzano, Italy
- Amsterdam UMC, Amsterdam, North Holland, Netherlands
- Guy's and St. Thomas' Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided